CLINICAL TRIAL: NCT07159867
Title: Frequency of Hypermobility-Related Problems in Patients With Anorexia Nervosa
Status: Not yet recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Elke Schubert Hjalmarsson, Dr, Vastra Gotaland Region
Other Study IDs: 2023-00568-01
Record Dates: First submitted 2025-08-21; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Anorexia Nervosa, Atypical; Anorexia Nervosa
Keywords: Anorexia nervosa; Joint hypermobility; Pain; Temporomandibular joint
MeSH Terms: conditions — Anorexia Nervosa; Joint Instability; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Female patients diagnosed with Anorexia Nervosa or Atypical Anorexia Nervosa, aged 13-25 years.

SUMMARY:
The purpose of this study is to examine the frequense of generalized hypermobility and pain in patients with Anorexia Nervosa. The study further explores two main questions: (1) whether generalized hypermobility may be an explanatory factor for pain in some patients with Anorexia Nervosa, and (2) whether temporomandibular joint problems (such as instability, pain, difficulties opening the mouth, locking, or clicking) contribute to eating difficulties in certain individuals with Anorexia Nervosa.

DETAILED DESCRIPTION:
Patients with eating disorder diagnosis Anorexia Nervosa, who are either currently in treatment or awaiting treatment at the Eating Disorders Center for children and young adults in Gothenburg, will be invited to participate in the study. During a single examination session, the patient's joints will be assessed to determine whether generalized hypermobility is present. At the same visit, the patient will answer questions regarding possible bodily pain and any temporomandibular joint problems. Joint mobility will be examined and assessed by a physiotherapist at the clinic. The examination follows a standardized protocol for assessing joint mobility and includes the assessment of nine specified joints.

ELIGIBILITY:
Inclusion Criteria:

Female patients Aged 13-25 years

Diagnosed with:

* Anorexia Nervosa (ICD-10 F50.0), or
* Atypical Anorexia Nervosa (ICD-10 F50.1)
* Currently receiving treatment or scheduled to receive treatment

Exclusion Criteria:

* Severe cognitive impairment
* Insufficient Swedish language skills that make it impossible to provide informed consent and prevent answering study questions
* Pregnancy and up to one year postpartum

Ages: 13 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients at the Eating Disorders Center for Children and Young Adults in Gothenburg.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Joint hypermobility | One-time assessment at baseline (Day 0, at the inclusion visit).
  Joint mobility will be assessed according to the Beighton score using a goniometer.
5-part questionnaire | One-time questionnaire at baseline (Day 0, after clinical examination).
  Participants over the age of 18 will also complete the 5-part questionnaire regarding historical hypermobility.

SECONDARY OUTCOMES:
Joint pain | One-time questionnaire at baseline (Day 0, after clinical examination).
  The Numeric Rating Scale (NRS) is a self-assessment tool used to describe the patient's perceived pain intensity. The patient marks the intensity on a line with eleven points, ranging from 0 to 10. The endpoints represent 0 = 'no pain' and 10 = 'worst imaginable pain.'
Temporomandibular joint problems | One-time questionnaire at baseline (Day 0, after clinical examination).
  Screening questions regarding temporomandibular joint problems. The short version of the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) classification system will be used.
Pain drawing | One-time questionnaire at baseline (Day 0, after clinical examination).
  Participant marks areas of perceived pain on a schematic human body figure.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Silvias Children´s Hospital, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No